CLINICAL TRIAL: NCT02344719
Title: The Effect of Oral Taurine on Portal Hemodynamics in Patients With Advanced
Brief Title: Effect of Taurine on Portal Hemodynamics in Patients With Advanced Liver Cirrhosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Arnulf Ferlitsch, MD, Assoz. Prof. Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2010-020880-19
Record Dates: First submitted 2015-01-12; First posted 2015-01-26 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Cirrhosis; Portal Hypertension
Keywords: cirrhosis; portal hypertension; taurin
MeSH Terms: conditions — Fibrosis; Hypertension, Portal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 6 capsules Taurin per day (Active Comparator): After baseline HVPG (Hepatic Venous Pressure Measurement)patients take 6x1g capsules of GMP produced Taurin per day, on day 28, after intake of the 6x1g Taurin capsules, HVPG measurement will be repeated.
  Interventions: Drug: Taurin 6g per day per oral for 28 days; Procedure: HVPG Measurement baseline; Procedure: HVPG Measurement day 28
- 6 capsuless placebo per day (Placebo Comparator): After baseline HVPG measurement patients take 6x1g capsules of placebo per day, on day 28, after intake of the 6x1g placebo capsules, HVPG measurement will be repeated.
  Interventions: Procedure: HVPG Measurement baseline; Procedure: HVPG Measurement day 28; Drug: Placebo 6g per day per oral for 28 days

INTERVENTIONS:
Drug: Taurin 6g per day per oral for 28 days — Taurin 6g per day per oral for 28 days
  Other Names: Taurin
  Arms: 6 capsules Taurin per day
Procedure: HVPG Measurement baseline — On day 1 (baseline) and day 28 HVPG measurement will be performed
  Other Names: HVPG
Procedure: HVPG Measurement day 28 — On day 1 (baseline) and day 28 HVPG measurement will be performed
  Other Names: HVPG
Drug: Placebo 6g per day per oral for 28 days — Placebo to Taurin 6g per day per oral for 28 days
  Arms: 6 capsuless placebo per day

SUMMARY:
The investigators want to analyze the effect of Taurin on portal hemodynamics in patients with advanced liver cirrhosis.

DETAILED DESCRIPTION:
28 days of 6 grams Taurine versus Placebo (randomization 1:1).

ELIGIBILITY:
Inclusion Criteria:

* Patients (male and female) aged older than 18 years with advanced liver cirrhosis (Child's Grade B and Child's Grade C), regardless of the disease origin (viral, alcoholic, idiopathic), who are scheduled for hepatic hemodynamic investigation
* Negative pregnancy test of women with childbearing potential
* Patient without beta blocker therapy: due to: intolerance of the medication, preexisting contraindication against beta blocker therapy, endoscopic band ligation as prophylaxis

Exclusion Criteria:

* History of variceal bleeding without endoscopic band ligation
* History of endoscopically diagnosed large varices with red spots without previous bleeding and without endoscopic band ligation
* HVPG < 10 mmHg
* HVPG > 20 mmHg and varices, unless ligated and treated in an eradication program within 6 months
* Beta Blocker therapy
* History of hypersensitivity to the trial drugs and contrast agent or to drugs with similar chemical structure
* Treatment with vasoactive or non-steroidal anti-inflammatory drugs or systematic antibiotics one week before the study
* Exclusion criteria for hepatic hemodynamic investigation
* Cardiac, renal or respiratory failure
* Previous surgical or transjugular intrahepatic portosystemic shunt
* Breast-feeding or pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-10; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
HVPG change in mmHg after 28 days with Taurin 6g or placebo | 28 days
  To investigate the response to 6g taurine p.o. for 28 days on the hepatic venous pressure gradient

CONTACTS AND LOCATIONS:
Overall Officials: Arnulf Ferlitsch, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Dept. of Internal Medicine III, Gastroenterology and Hepatology, Medical University of Vienna, Vienna, Austria